CLINICAL TRIAL: NCT04246944
Title: Induced Membrane Properties in Children and Adults
Acronym: EMIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2018_843_0041
Record Dates: First submitted 2020-01-17; First posted 2020-01-29 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Bone Loss; Surgery
Keywords: induced membrane; critical size defect
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: harvesting induced membrane — The induced membrane will be harvested during the second step of the bone reconstruction.

SUMMARY:
Bone reconstruction in critical sized defect (CSD) remains a real challenge in orthopedic surgery in children and adults. The Masquelet technique is an innovative therapeutic technique, which offers a bone reconstruction in two steps, by the formation of an induced membrane (IM) around a polymethylmethacrylate (PMMA) spacer placed into the bone defect. After, PMMA removal, the cavity is filled with corticocancellous graft allowing bone healing. Up to date, all angiogenesis and osteogenic properties of IM remain unknown. The purpose of this study is to characterize angiogenesis and osteogenic properties of IM in children and adults.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated at CHU Amiens-Picardie for bone critical sized defect treated using the induced membrane reconstruction technique.
* patients from 9 months to 60 years old

Exclusion Criteria:

* Patients managed by another reconstruction technique for critical sized defect
* Patients under guardianship, curators or deprived of liberty.
* Pregnant and nursing women.
* Patients who refused to participate in the study and to sign informed consent.

Ages: 9 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Measure of the BMP2 concentration of the induced membrane by immunodetection | one year (one year from day of surgery)
  Measure of the osteogenic property of the induced membrane will be made after harvesting the induced membrane

SECONDARY OUTCOMES:
BMP2 concentration of the induced membrane implanted in adults measured by immunodetection | one year (one year from day of surgery)
  measurement of osteogenic property of the induced membrane in adults
BMP2 concentration of the induced membrane implanted in children measured by immunodetection | one year (one year from day of surgery)
  measurement of osteogenic property of the induced membrane in children

CONTACTS AND LOCATIONS:
Overall Officials: Céline Klein, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No